CLINICAL TRIAL: NCT00022854
Title: Outcomes After ACL Reconstruction: The Effect of Femoral Nerve Block Analgesia
Brief Title: Pain Relief Results After Anterior Cruciate Ligament (ACL) Reconstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K23AR047631 (NIH); K23AR047631 (NIH); NIAMS-066
Record Dates: First submitted 2001-08-14; First posted 2001-08-16 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: ACL; Nerve block; Knee; Outcome survey; Anesthesia; Analgesia; Pain
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Agnosia; Pain | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator)
  Interventions: Procedure: Saline (control) injection into femoral nerve envelope
- 2 (Experimental): Nerve block bolus with 30 mL levobupivacaine 0.25%, followed by continuous saline infusion
  Interventions: Procedure: Single-injection femoral nerve block
- 3 (Experimental): Nerve block bolus with 30 mL levobupivacaine 0.25%, followed by continuous levobupivacaine infusion of 5 mL/hr for 50 hr
  Interventions: Procedure: Femoral nerve block 60-hour continuous injection

INTERVENTIONS:
Procedure: Single-injection femoral nerve block — Nerve block bolus with 30 mL levobupivacaine 0.25%, followed by continuous saline infusion
  Arms: 2
Procedure: Femoral nerve block 60-hour continuous injection — Nerve block bolus with 30 mL levobupivacaine 0.25%, followed by continuous infusion (5 mL/hr for 50 hours) of 0.25% levobupivacaine
  Arms: 3
Procedure: Saline (control) injection into femoral nerve envelope — Nerve block bolus with 30 mL saline, followed by continuous saline infusion
  Arms: 1

SUMMARY:
Anterior cruciate ligament (ACL) reconstruction is surgery that is done to repair a damaged ligament in the knee. In this study we will look at whether the femoral nerve block, a commonly used method for pain relief after ACL reconstruction, affects the way patients feel after surgery. We will study recovery during the first week after surgery and also 3-12 weeks after surgery. We will give all patients spinal anesthesia. Some patients will also receive a continuous femoral nerve block for 2 days, or by a single injection. We predict that patients who received the nerve block will have significantly improved pain results, compared to patients who did not receive the nerve block.

DETAILED DESCRIPTION:
In this project, we will measure outcomes of anesthesia and pain management for common orthopedic procedures. The influence of nerve block pain management on outcomes after outpatient anterior cruciate ligament (ACL) reconstruction has not been studied, especially the patient's potential to return to societal productivity during the first week after surgery. Therefore, we have designed a randomized clinical trial to study the role of nerve block pain management techniques on patient outcomes during the first week after surgery and on recovery 3-12 weeks after surgery. Our hypothesis is that patients undergoing nerve block analgesia will manifest better self-reported recovery outcomes, physical function outcomes, and objective measures of neuromuscular function.

We will give consenting patients (n=270) undergoing ACL reconstruction conventional spinal anesthesia and will randomize them to receive femoral nerve block analgesia with either a single injection, a continuous infusion for 2 days, or saline placebo. We will use goniometry to test postoperative range of motion in extension to determine whether the quadriceps femoris torque output is impaired. We will compare patient-reported recovery outcomes across treatment groups using three validated health status measures suitable for daily assessment (Verbal Pain Score, SF-8, and the Quality of Recovery [from anesthesia, QoR-40] Score).

We aim to determine the quality of immediate recovery from anesthesia and the extent of reported pain. We will compare the effects of single injection and continuous infusion on femoral nerve analgesia to determine the better dosing strategy for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-65
* Undergoing ACL reconstruction at the University of Pittsburgh
* Agrees to spinal anesthesia and consents to one of the three nerve block interventions.
* Agrees to visit the University of Pittsburgh Center for Rehabilitation Services for postoperative physical therapy and rehabilitation (for standardized rehabilitation protocols)

Exclusion Criteria:

* Morbid obesity
* Chronic pain syndromes
* Opioid dependence
* Corticosteroid prescriptions
* Tricyclic antidepressant prescriptions
* Tramadol prescriptions
* Preexisting neuropathies
* Poorly controlled diabetes mellitus
* Poorly controlled anxiety disorders

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2001-05; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Pain scores during the first week after surgery | one week

SECONDARY OUTCOMES:
Side effects during the first week after surgery (nausea, vomiting, quality of sleep) | first week after surgery
Determine the "rebound pain score" after a nerve block wears off | first week after surgery
Skin reactions to the nerve block catehter dressing | first week after surgery
Risk of falling | first week after surgery
Validation of an 8-item outcome survey in comparison to a 40-item "gold standard" outcome survey | first week after surgery
Study staffing costs before and after the implementation of HIPAA | the 40 months of study recruitment
Patient-reported general health status, and patient-reported knee function, during the first 12 weeks after surgery | up to 12 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Brian A. Williams, MD, MBA, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Center for Sports Medicine, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Williams BA, Kentor ML, Williams JP, Figallo CM, Sigl JC, Anders JW, Bear TC, Tullock WC, Bennett CH, Harner CD, Fu FH. Process analysis in outpatient knee surgery: effects of regional and general anesthesia on anesthesia-controlled time. Anesthesiology. 2000 Aug;93(2):529-38. doi: 10.1097/00000542-200008000-00033. PMID 10910504
- [Background] Williams BA, Kentor ML, Williams JP, Vogt MT, DaPos SV, Harner CD, Fu FH. PACU bypass after outpatient knee surgery is associated with fewer unplanned hospital admissions but more phase II nursing interventions. Anesthesiology. 2002 Oct;97(4):981-8. doi: 10.1097/00000542-200210000-00034. PMID 12357168
- [Background] Williams BA, Kentor ML, Vogt MT, Williams JP, Chelly JE, Valalik S, Harner CD, Fu FH. Femoral-sciatic nerve blocks for complex outpatient knee surgery are associated with less postoperative pain before same-day discharge: a review of 1,200 consecutive cases from the period 1996-1999. Anesthesiology. 2003 May;98(5):1206-13. doi: 10.1097/00000542-200305000-00024. PMID 12717143
- [Background] Williams BA, Kentor ML, Vogt MT, Vogt WB, Coley KC, Williams JP, Roberts MS, Chelly JE, Harner CD, Fu FH. Economics of nerve block pain management after anterior cruciate ligament reconstruction: potential hospital cost savings via associated postanesthesia care unit bypass and same-day discharge. Anesthesiology. 2004 Mar;100(3):697-706. doi: 10.1097/00000542-200403000-00034. PMID 15108988
- [Result] Williams BA, Kentor ML, Vogt MT, Irrgang JJ, Bottegal MT, West RV, Harner CD, Fu FH, Williams JP. Reduction of verbal pain scores after anterior cruciate ligament reconstruction with 2-day continuous femoral nerve block: a randomized clinical trial. Anesthesiology. 2006 Feb;104(2):315-27. doi: 10.1097/00000542-200602000-00018. PMID 16436852
- [Result] Williams BA, Kentor ML, Irrgang JJ, Bottegal MT, Williams JP. Nausea, vomiting, sleep, and restfulness upon discharge home after outpatient anterior cruciate ligament reconstruction with regional anesthesia and multimodal analgesia/antiemesis. Reg Anesth Pain Med. 2007 May-Jun;32(3):193-202. doi: 10.1016/j.rapm.2006.12.002. PMID 17543813
- [Result] Williams BA, Bottegal MT, Kentor ML, Irrgang JJ, Williams JP. Rebound pain scores as a function of femoral nerve block duration after anterior cruciate ligament reconstruction: retrospective analysis of a prospective, randomized clinical trial. Reg Anesth Pain Med. 2007 May-Jun;32(3):186-92. doi: 10.1016/j.rapm.2006.10.011. PMID 17543812
- [Result] Bost JE, Williams BA, Bottegal MT, Dang Q, Rubio DM. The 8-item Short-Form Health Survey and the physical comfort composite score of the quality of recovery 40-item scale provide the most responsive assessments of pain, physical function, and mental function during the first 4 days after ambulatory knee surgery with regional anesthesia. Anesth Analg. 2007 Dec;105(6):1693-700, table of contents. doi: 10.1213/01.ane.0000287659.14893.65. PMID 18042869
- [Result] Williams BA, Kentor ML, Bottegal MT. The incidence of falls at home in patients with perineural femoral catheters: a retrospective summary of a randomized clinical trial. Anesth Analg. 2007 Apr;104(4):1002. doi: 10.1213/01.ane.0000256006.46703.7f. No abstract available. PMID 17377133
- [Result] Williams BA, Bolland MA, Orebaugh SL, Bottegal MT, Kentor ML. Skin reactions at the femoral perineural catheter insertion site: retrospective summary of a randomized clinical trial. Anesth Analg. 2007 May;104(5):1309-10. doi: 10.1213/01.ane.0000260353.11142.d4. No abstract available. PMID 17456710
- [Result] Williams BA, Bottegal MT, Francis KA, Irrgang JJ, Vogt MT. A post hoc analysis of research study staffing: budgetary effects of the Health Insurance Portability and Accountability Act on research staff work hours during a prospective, randomized clinical trial. Anesthesiology. 2007 Nov;107(5):860-1. doi: 10.1097/01.anes.0000287212.90397.6b. No abstract available. PMID 18073577